CLINICAL TRIAL: NCT00935675
Title: Double-blind, Placebo-controlled, Randomized Study of the Effectiveness of Escitalopram on Emotional Distress of Head and Neck Cancer Patients During Cancer Treatment
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: SARAH DAUCHY MD
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TADDOR; CSET 1388
Record Dates: First submitted 2009-07-07; First posted 2009-07-09 (Estimated); Last update posted 2009-09-02 (Estimated); Status verified 2009-07

CONDITIONS: Carcinomas
Keywords: Patients with head and neck squamous cell carcinomas; head and neck squamous cell carcinomas
MeSH Terms: conditions — Carcinoma; Squamous Cell Carcinoma of Head and Neck | interventions — Escitalopram

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Antidepressant treatment (Active Comparator)
  Interventions: Drug: Escitalopram
- Placebo (Placebo Comparator)
  Interventions: Drug: Escitalopram

INTERVENTIONS:
Drug: Escitalopram — Escitalopram 10 mg once a day

SUMMARY:
Evaluation of the effectiveness of escitalopram on depressive symptoms after 3 months in patients with head and neck squamous cell carcinomas (oral cavity, larynx, oropharynx and hypopharynx) and with an HADS total score > 11

ELIGIBILITY:
Inclusion Criteria:

1. Head and neck squamous cell carcinomas, stage I to IVb
2. First-line curative cancer therapy : surgery and/or brachytherapy and/or chemotherapy
3. HADS- T >11
4. Aged 18 to 75 yo, written consent required
5. OMS>2

Exclusion Criteria:

1. Palliative care
2. Previous head and neck cancer
3. Bipolar disorder or schizophrenia
4. Severe major depressive disorder (DSM-IV TR)
5. Expressed suicidal ideation
6. Severe untreated organic disorder, especially acute infectious disorder
7. ASAT/ALAT > 3N
8. Clearance of creatinin < 30 ml/mn
9. Hyponatremia
10. Antecedent of delirium tremens or acute alcohol withdrawal disorder
11. Antecedent of upper gastro-intestinal bleeding
12. Antecedent of toxicity or inefficacy of a previous treatment with escitalopram
13. Unauthorized treatments :- Antidepressant or antiepileptic (clonazepam authorized)- Hypnotic except zolpidem - Anxiolytic except clonazepam, clorazepate or diazepam- bupropion or varenicline
14. Pregnancy or lactation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the effectiveness of escitalopram on depressive symptoms after 3 months | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Gustave Roussy, Villejuif, France

REFERENCES:
- [Derived] Vita G, Compri B, Matcham F, Barbui C, Ostuzzi G. Antidepressants for the treatment of depression in people with cancer. Cochrane Database Syst Rev. 2023 Mar 31;3(3):CD011006. doi: 10.1002/14651858.CD011006.pub4. PMID 36999619
- See also: Related Info — http://www.igr.fr/